CLINICAL TRIAL: NCT01278563
Title: A Randomized Controlled Trial to Investigate the Impact of a Low Glycemic Index (GI) Diet on Body Mass Index and Obesity Related Cardiovascular and Hormonal Factors in Chinese Adolescents
Brief Title: A Trial to Investigate the Impact of a Low Glycemic Index (GI) Diet on Body Mass Index and Obesity Related Cardiovascular and Hormonal Factors in Chinese Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Alice Pik Shan KONG, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGC467410
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Adolescence Obesity
Keywords: Low Glycemic Index Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Low glycemic index diet — dietitian interview and counselling for the low glycemic index diet group

SUMMARY:
Epidemiological studies suggest a role for a low glycemic index (GI) diet in the management of obesity and associated metabolic risks including diabetes. However, evidence from long-term, randomized controlled trials exploring the relationship between low GI diet, weight reduction and glycemia, particularly in children and adolescents, is lacking. Modern food-processing technology has produced many food products with high GI which may contribute to the burgeoning epidemic of obesity worldwide. Since dietary habits are shaped in early life, adolescence is a critical period to educate our young people to acquire a healthy eating habit to prevent obesity.

The investigators hypothesized that, in Chinese adolescents, low GI diet results in greater reduction in body mass index and body fat percentage, enhanced insulin sensitivity and favorable changes of cardiometabolic risk factors compared to conventional diet after 12 months of intervention.

This study is a randomized controlled trial of a low GI (<55) versus conventional Chinese diet (GI>/=70) in adolescents (12-month intervention followed by a 6-month observational period) to study; 1) the changes in body mass index and obesity associated changes in cardiometabolic profile; 2) the underlying hormonal factors associated with these changes.

DETAILED DESCRIPTION:
This is a 12-month randomized controlled dietary interventional trial followed by a 6-month observational period. The objectives of this study include:

1. To study changes of body mass index, body fat percentage, insulin secretion, insulin resistance and obesity associated cardiometabolic factors;
2. To explore underlying neurohormonal mechanisms associated with these changes in both short- and long-term.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 and 18 years (inclusive)
* Male or female of Chinese ethnicity
* Body mass index >/= 95th percentile of Hong Kong local age- and sex-specific reference
* No major medical illness
* Not on any chronic medications
* Post-pubertal as ascertained by clinical assessment by endocrinologist
* Willingness to give written informed consent by participants and his/her parents/guardian

Exclusion criteria:

* Concurrent participation in any clinical trial, dietary intervention or weight loss program
* Concomitant intake of weight reducing agent
* Active and uncontrolled endocrine diseases including hypo- or hyperthyroidism, Cushing's syndrome, diabetes mellitus, etc.
* Significant renal impairment, defined as serum creatinine >150 umol/L and/or estimated glomerular filtration rate <60ml/min/1.73m2
* Significant liver impairment, defined as >2 times upper limit of alanine aminotransferase and asparate aminotransferase levels
* Gastrointestinal problems that would prevent them from following the test diets
* Active malignant disease
* Pregnant or lactating
* Any medical illness or condition including known non-compliance, as judged by the investigators as ineligible to participate the study

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
body mass index | change from baseline to 12 months
  body mass index= body weight (kg) divided by square of body height (m2)

SECONDARY OUTCOMES:
other parameters of body composition | change from baseline to 12 months
  1. waist circumference
  2. body fat percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Centre, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Kong AP, Choi KC, Chan RS, Lok K, Ozaki R, Li AM, Ho CS, Chan MH, Sea M, Henry CJ, Chan JC, Woo J. A randomized controlled trial to investigate the impact of a low glycemic index (GI) diet on body mass index in obese adolescents. BMC Public Health. 2014 Feb 19;14:180. doi: 10.1186/1471-2458-14-180. PMID 24552366